CLINICAL TRIAL: NCT04617626
Title: REACH Côte d'Ivoire: Feasibility and Acceptability of Integrating Mass Distribution of Azithromycin to Children 1-11 Months Into a Trachoma Mass Drug Administration Campaign to Reduce Child Mortality
Brief Title: Resiliency Through Azithromycin for Children (REACH), Côte d'Ivoire
Acronym: REACH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FHI 360 (Other)
Collaborators: National Program for the Fight Against Neglected Tropical Diseases, Côte d'Ivoire (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 1575564
Record Dates: First submitted 2020-10-16; First posted 2020-11-05 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Child Mortality; Azithromycin
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Azithromycin (Other): All children ages 1 to 5 months in the targeted health district will be offered a single dose of azithromycin suspension dosed at 20 mg per kg of weight in place of the standard tetracycline ointment, during a mass drug administration targeting trachoma prevention and treatment. All children ages 6 months and older, and all adults already receive the single dose of azithromycin during the MDA event. For this pilot study, single dose of azithromycin is being extended to include the 1 to 5 month old population as well.
  Interventions: Drug: Azithromycin

INTERVENTIONS:
Drug: Azithromycin — Single dose of azithromycin suspension

SUMMARY:
The aim of the study is to gather preliminary evidence on the operational feasibility and acceptability of integrating bi-annual mass drug administration (MDA) of single-dose azithromycin for children ages 1 to 11 months in high child mortality settings in Côte. The cross-sectional study will be carried out in conjunction with a single trachoma MDA in selected villages within one health district. Data on feasibility and acceptability will be collected through three main activities:

1. Analyses of existing routine monitoring, process, and adverse drug reaction data from the trachoma MDA platform into which the pilot activities are being integrated
2. A cross-sectional, post-MDA coverage survey
3. Qualitative data collection among targeting parents or primary caregivers of children ages 1 to 11 months in the pilot districts, and district-level MDA implementers, regarding the proposed azithromycin program.

DETAILED DESCRIPTION:
Purpose: The aim of the study is to gather preliminary evidence on the operational feasibility and acceptability of integrating bi-annual mass drug administration (MDA) of single-dose azithromycin for children ages 1 to 11 months in high child mortality settings in Côte d'Ivoire into the existing trachoma MDA platform to inform large scale implementation.

Design: The cross-sectional study will be carried out in conjunction with a single trachoma MDA in selected villages within one health district. Data on feasibility and acceptability will be collected through three main activities:

1. Analyses of existing routine monitoring, process, and adverse drug reaction data from the trachoma MDA platform into which the pilot activities are being integrated
2. A cross-sectional, post-MDA coverage survey
3. Qualitative data collection among targeting parents or primary caregivers of children ages 1 to 11 months in the pilot districts, and district-level MDA implementers, regarding the proposed azithromycin program.

Population: For expanded use of azithromycin: Infants ages 1 to 5 months who reside in one pilot district in high under-5 years child mortality regions in Côte d'Ivoire (approximately 2,800 to be enrolled).

Post-MDA coverage survey and interviews for acceptability: Parents/primary caregivers of infants aged 1 to 11 months who reside in the two pilot districts will be targeted for the post-MDA coverage survey and in-depth interviews (n=up to 24) to explore acceptability (approximately 275 to be enrolled).

Feasibility and acceptability from implementers' perspectives: Focus group discussions will target community-based drug distributors (CDDs) and in-depth interviews will target CDD supervisors, both to explore operational feasibility. (A maximum of 48 CDDs and 12 CDD supervisors approximately) Pilot Site : Boundiali Health District in Bagoué Region, among the high under-5 child mortality regions in Côte d'Ivoire.

Duration: Planning - 6 months; Training and implementation of the pilot intervention - 3 weeks; Post-MDA research - 1 month; Data analysis and reporting - 2 months.

Objectives: The study is designed to:

1. Examine the extent to which activities are carried out as planned (fidelity) during the pilot implementation and the factors that affect the processes and results.
2. Estimate coverage of the intervention's target population (1 to 11 month-olds) with azithromycin in pilot districts.
3. Assess the level of understanding and acceptability of the strategy among those involved in implementation and among the parents/primary caregivers of children targeted by the intervention.
4. Document challenges to implementation and costs of the pilot activity to make recommendations for scale-up.

Endpoints: A final pilot activity report summarizing findings including recommended approaches for scale-up, will be developed after results are shared with the REACH technical working group to inform guidance on scale-up.

ELIGIBILITY:
For expanded azithromycin access during the MDA

Inclusion Criteria:

* Child aged 1 month (at least 30 days) to less than 6 months at the beginning of the week of the MDA intervention
* Resident in study communities

Exclusion Criteria:

* Children below 3.0 kg
* Appears severely ill at the time of the MDA (per the CDD's assessment)
* Unable to swallow liquid delivered through a needle-less syringe because of physical limitations
* Known allergy to macrolides, including azithromycin, based on the primary caregiver's report of prior adverse reaction to medication likely to be a macrolide

Ages: 1 Month to 5 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1735 (Actual)
Dates: Start 2020-11-20 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Proportion of children 1 to 11 months reached with single-dose azithromycin | 1 week
  The proportion of children 1 to 11 months of age who receive a single dose of azithromycin during the MDA in the target health district.

CONTACTS AND LOCATIONS:
Locations (1):
- Boundiali Health District, Boundiali, Savanes District, Côte d’Ivoire

IPD SHARING:
Plan to Share IPD: Yes
De-identified data from the study survey will be posted to a data sharing site, such as Harvard Dataverse, upon conclusion of the study.
Supporting Information: Study Protocol, ICF
Time Frame: To be made available indefinitely after Feb. 28, 2020.

REFERENCES:
- [Derived] Dulli L, Toure F, Mama AD, Evens E, Murray K, Dje NN, Kone S, Sadate-Ngatchou P, Bovary A, Eichleay M, Jean-Baptiste M, Meite A. Feasibility and acceptability of integrating mass distribution of azithromycin to children 1-11 months into a trachoma mass drug administration campaign to reduce child mortality in Cote d'Ivoire. PLOS Glob Public Health. 2024 Jul 10;4(7):e0003426. doi: 10.1371/journal.pgph.0003426. eCollection 2024. PMID 38985785